CLINICAL TRIAL: NCT03099512
Title: The Effects of Foot Exercises on Pain, Biomechanical Characteristics and Functionality of Lower Extremity in Patients With Patellofemoral Pain
Brief Title: The Foot Exercises in Patellofemoral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Pınar Kısacık, Research Asistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 17/168
Record Dates: First submitted 2017-03-18; First posted 2017-04-04 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Patellofemoral Pain Syndrome; Anterior Knee Pain Syndrome; Pronation Deformity of the Foot; Exercise; Pain; Biomechanics; Functionality
Keywords: Patellofemoral pain; foot deformity; foot pronation; short foot exercise
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Motor Activity; Pain; Foot Deformities | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ex+SFE Group (Experimental): Individuals in this group who will perform exercises for knee and also short foot exercise
  Interventions: Other: SFE; Other: Exercise
- Ex Group (Active Comparator): Individuals in this group who will perform exercises for knee only
  Interventions: Other: Exercise

INTERVENTIONS:
Other: SFE — The 'short foot exercise' has been described as a means to isolate contraction of the plantar intrinsic muscles.
  Arms: Ex+SFE Group
Other: Exercise — Exercises which improves muscle strength, ROM...

SUMMARY:
The purpose of this study is to investigate the additional effects of Short Foot Exercises on pain, biomechanical characteristics and functionality of lower extremity in patients with patellofemoral pain.

ELIGIBILITY:
Inclusion Criteria:

* aged between 25-60
* diagnosed as patellofemoral pain syndrome

Exclusion Criteria:

* Pregnancy
* Having walking disability
* Having a trauma, knee surgery or other arthritis

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Change from baseline pain at 6th week
  Asked for expression of pain

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Kısacık, Principal Investigator — Hacettepe University
Locations (1):
- Pınar Kısacık, Ankara, Turkey (Türkiye)